CLINICAL TRIAL: NCT03267615
Title: VICIS - Vienna Cirrhosis Study
Acronym: VICIS
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Reiberger, Univ.-Prof. Priv-Doz. Dr., Medical University of Vienna
Other Study IDs: VICIS
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Ascites; Variceal Hemorrhage; Hepatic Encephalopathy
Keywords: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Ascites; Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Plasma, Serum, Urine, Stool, GI mucosa biopsies, ascitic fluid, liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with advanced chronic liver diseases treated at the Vienna General Hospital of the Medical University of Vienna will be offered to participate in this prospective observational trial - including an optional participation in a biobank.

Clinical parameters and laboratory parameters will be recorded for all patients and patients will undergo a regular follow-up schedule with clinical visits at the Vienna General Hospital.

This study is linked to a biobank with serum/plasma, ascitic fluid, urine, GI tract mucosal biopsies, liver biopsies and stool collected from the study participants.

DETAILED DESCRIPTION:
Patients with advanced chronic liver disease (ACLD) as evident by HVPG>5mmHg or liver biopsy showing F3/F4 fibrosis or as suggested by liver stiffness measurement (LSM) ≥10kPa can be included in the VICIS study. Most patients will be recruited on the day of HVPG measurement performed for screening of clinically significant portal hypertension (CSPH) or on the day of upper GI endoscopy for screening for the presence of varices. Next to the detailed characterization of patients by epidemiologic, clinical and laboratory parameters, the degree of portal hypertension will be assessed by HVPG, liver (LSM) and spleen (SSM) stiffness will be assessed by transient elastography, the presence of ascites, splenomegaly, portosystemic collaterals, PVT and liver lesions will be assessed by ultrasound and optionally cross-sectional imaging.

In addition, patients will be asked to (optionally) participate in biobank sampling including serum/plasma, ascitic fluid, urine, GI tract mucosal biopsies, stool, liver biopsies and stool. All patients recruited in the VICIS study will be prospectively followed every 3 months (decompenated ACLD) or every 6 months (compensated ACLD) patients with clinical visits at the Cirrhosis Outpatient Clinic at the Vienna General Hospital. These assessments include a detailed assessment of risk factors (such as a structured interview of alcohol consumption), the recording of decompensating events (such as ascites, hepatic encephalopathy, variceal bleeding), screening for PVT and HCC, recording of medications and other clinically-relevant information.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <100 years
* Diagnosis of advanced chronic liver disease (by liver stiffness ≥10kPa, HVPG>5mmHg or Histology F3/F4)
* Written informed consent

Exclusion Criteria:

* Withdrawal of written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced chronic liver disease diagnosed and/or treated at the Medical University of Vienna will be screened for inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival | 01/FEB/2017 - 31/DECEMBER/2027
  Time from inclusion to death or liver transplantation

SECONDARY OUTCOMES:
Decompensation-free survival | 01/FEB/2017 - 31/DECEMBER/2027
  Time from inclusion to decompensation, death or liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reiberger, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kramer G, Simbrunner B, Jachs M, Balcar L, Hofer BS, Dominik N, Hartl L, Schwarz M, Semmler G, Sebesta C, Thone P, Geisselbrecht S, Maasoumy B, Alvarez E, McCoy MS, Petrenko O, Reinis J, Schwabl P, Stattermayer AF, Trauner M, Mandorfer M, Reiberger T. Blood-based Vienna 3P/5P risk models accurately predict first hepatic decompensation in compensated advanced chronic liver disease. JHEP Rep. 2025 Oct 17;8(2):101642. doi: 10.1016/j.jhepr.2025.101642. eCollection 2026 Feb. PMID 41551411
- [Derived] Jachs M, Carvalho T, Simbrunner B, Semmler G, Hartl L, Balcar L, Hofer BS, Thone P, Dominik N, Kramer G, Sebesta C, Schwarz M, Bauer D, Stattermayer AF, Pinter M, Trauner M, Reiberger T, Mandorfer M. Indocyanine Green Clearance Correlates With Biomarkers Reflecting Key Disease-Driving Mechanisms in Advanced Chronic Liver Disease and Predicts Acute-on-Chronic Liver Failure and Death. Aliment Pharmacol Ther. 2025 Nov 5. doi: 10.1111/apt.70447. Online ahead of print. PMID 41194563
- [Derived] Simbrunner B, Villesen IF, Semmler G, Balcar L, Kramer G, Almeida Calvao J, Hofer BS, Jachs M, Hartl L, Maurer J, Scheiner B, Zinober K, Marculescu R, Trauner M, Karsdal M, Reiberger T, Mandorfer M, Leeming DJ. Biomarkers of Extracellular Matrix Remodelling Are Linked to Severity and Outcome of Advanced Chronic Liver Disease. Aliment Pharmacol Ther. 2025 Oct 12. doi: 10.1111/apt.70407. Online ahead of print. PMID 41077886
- [Derived] Dominik N, Simbrunner B, Scheiner B, Schwarz M, Hartl L, Jachs M, Balcar L, Semmler G, Kramer G, Sebesta C, Trauner M, Pinter M, Mandorfer M, Reiberger T, Hofer BS. Smoking Aggravates Inflammation, Fibrogenesis, Angiogenesis and Cancer Risk in Patients With Cirrhosis. Liver Int. 2025 Oct;45(10):e70314. doi: 10.1111/liv.70314. PMID 40899194
- [Derived] Hofer BS, Simbrunner B, Konigshofer P, Brusilovskaya K, Petrenko O, Taru V, Sorz-Nechay T, Zinober K, Regnat K, Semmler G, Lackner C, Trauner M, Mandorfer M, Schwabl P, Reiberger T. Inflammation remains a dynamic component of portal hypertension in regressive alcohol-related cirrhosis. United European Gastroenterol J. 2025 Apr;13(3):317-329. doi: 10.1002/ueg2.12643. Epub 2024 Dec 21. PMID 39708052
- [Derived] Simbrunner B, Hofer BS, Schwabl P, Zinober K, Petrenko O, Fuchs C, Semmler G, Marculescu R, Mandorfer M, Datz C, Trauner M, Reiberger T. FXR-FGF19 signaling in the gut-liver axis is dysregulated in patients with cirrhosis and correlates with impaired intestinal defence. Hepatol Int. 2024 Jun;18(3):929-942. doi: 10.1007/s12072-023-10636-4. Epub 2024 Feb 8. PMID 38332428
- [Derived] Hartl L, Simbrunner B, Jachs M, Wolf P, Bauer DJM, Scheiner B, Balcar L, Semmler G, Schwarz M, Marculescu R, Dannenberg V, Trauner M, Mandorfer M, Reiberger T. Lower free triiodothyronine (fT3) levels in cirrhosis are linked to systemic inflammation, higher risk of acute-on-chronic liver failure, and mortality. JHEP Rep. 2023 Nov 1;6(1):100954. doi: 10.1016/j.jhepr.2023.100954. eCollection 2024 Jan. PMID 38125301
- [Derived] Simbrunner B, Villesen IF, Scheiner B, Paternostro R, Schwabl P, Stattermayer AF, Marculescu R, Pinter M, Quehenberger P, Trauner M, Karsdal M, Lisman T, Reiberger T, Leeming DJ, Mandorfer M. Von Willebrand factor processing in patients with advanced chronic liver disease and its relation to portal hypertension and clinical outcome. Hepatol Int. 2023 Dec;17(6):1532-1544. doi: 10.1007/s12072-023-10577-y. Epub 2023 Aug 21. PMID 37605068
- [Derived] Hartl L, Simbrunner B, Jachs M, Wolf P, Bauer DJM, Scheiner B, Balcar L, Semmler G, Schwarz M, Marculescu R, Trauner M, Mandorfer M, Reiberger T. An impaired pituitary-adrenal signalling axis in stable cirrhosis is linked to worse prognosis. JHEP Rep. 2023 May 11;5(8):100789. doi: 10.1016/j.jhepr.2023.100789. eCollection 2023 Aug. PMID 37484210
- [Derived] Hofer BS, Simbrunner B, Hartl L, Jachs M, Balcar L, Paternostro R, Schwabl P, Semmler G, Scheiner B, Trauner M, Mandorfer M, Reiberger T. Hepatic recompensation according to Baveno VII criteria is linked to a significant survival benefit in decompensated alcohol-related cirrhosis. Liver Int. 2023 Oct;43(10):2220-2231. doi: 10.1111/liv.15676. Epub 2023 Jul 20. PMID 37469291
- [Derived] Simbrunner B, Hartl L, Jachs M, Bauer DJM, Scheiner B, Hofer BS, Stattermayer AF, Marculescu R, Trauner M, Mandorfer M, Reiberger T. Dysregulated biomarkers of innate and adaptive immunity predict infections and disease progression in cirrhosis. JHEP Rep. 2023 Feb 24;5(5):100712. doi: 10.1016/j.jhepr.2023.100712. eCollection 2023 May. PMID 37035457
- [Derived] Simbrunner B, Caparros E, Neuwirth T, Schwabl P, Konigshofer P, Bauer D, Marculescu R, Trauner M, Scheiner B, Stary G, Mandorfer M, Reiberger T, Frances R. Bacterial translocation occurs early in cirrhosis and triggers a selective inflammatory response. Hepatol Int. 2023 Aug;17(4):1045-1056. doi: 10.1007/s12072-023-10496-y. Epub 2023 Mar 7. PMID 36881247
- [Derived] Balcar L, Krawanja J, Scheiner B, Paternostro R, Simbrunner B, Semmler G, Jachs M, Hartl L, Stattermayer AF, Schwabl P, Pinter M, Szekeres T, Trauner M, Reiberger T, Mandorfer M. Impact of ammonia levels on outcome in clinically stable outpatients with advanced chronic liver disease. JHEP Rep. 2023 Jan 23;5(4):100682. doi: 10.1016/j.jhepr.2023.100682. eCollection 2023 Apr. PMID 36873421
- [Derived] Hofer BS, Simbrunner B, Hartl L, Jachs M, Bauer DJM, Balcar L, Paternostro R, Schwabl P, Semmler G, Scheiner B, Staettermayer AF, Trauner M, Mandorfer M, Reiberger T. Alcohol Abstinence Improves Prognosis Across All Stages of Portal Hypertension in Alcohol-Related Cirrhosis. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2308-2317.e7. doi: 10.1016/j.cgh.2022.11.033. Epub 2022 Dec 5. PMID 36481475
- [Derived] Reinis J, Petrenko O, Simbrunner B, Hofer BS, Schepis F, Scoppettuolo M, Saltini D, Indulti F, Guasconi T, Albillos A, Tellez L, Villanueva C, Brujats A, Garcia-Pagan JC, Perez-Campuzano V, Hernandez-Gea V, Rautou PE, Moga L, Vanwolleghem T, Kwanten WJ, Francque S, Trebicka J, Gu W, Ferstl PG, Gluud LL, Bendtsen F, Moller S, Kubicek S, Mandorfer M, Reiberger T. Assessment of portal hypertension severity using machine learning models in patients with compensated cirrhosis. J Hepatol. 2023 Feb;78(2):390-400. doi: 10.1016/j.jhep.2022.09.012. Epub 2022 Sep 22. PMID 36152767
- [Derived] Simbrunner B, Villesen IF, Konigshofer P, Scheiner B, Bauer D, Paternostro R, Schwabl P, Timelthaler G, Ramazanova D, Woran K, Stift J, Eigenbauer E, Stattermayer AF, Marculescu R, Pinter M, Moller S, Trauner M, Karsdal M, Leeming DJ, Reiberger T, Mandorfer M. Systemic inflammation is linked to liver fibrogenesis in patients with advanced chronic liver disease. Liver Int. 2022 Nov;42(11):2501-2512. doi: 10.1111/liv.15365. Epub 2022 Aug 25. PMID 35822301
- [Derived] Hofer BS, Simbrunner B, Bauer DJM, Paternostro R, Schwabl P, Scheiner B, Semmler G, Hartl L, Jachs M, Datterl B, Staettermayer AF, Trauner M, Mandorfer M, Reiberger T. Acute hemodynamic response to propranolol predicts bleeding and nonbleeding decompensation in patients with cirrhosis. Hepatol Commun. 2022 Sep;6(9):2569-2580. doi: 10.1002/hep4.2021. Epub 2022 Jul 8. PMID 35808889
- [Derived] Scheiner B, Balcar L, Nussbaumer RJ, Weinzierl J, Paternostro R, Simbrunner B, Hartl L, Jachs M, Bauer D, Stattermayer AF, Semmler G, Pinter M, Ay C, Quehenberger P, Trauner M, Reiberger T, Lisman T, Mandorfer M. Factor VIII/protein C ratio independently predicts liver-related events but does not indicate a hypercoagulable state in ACLD. J Hepatol. 2022 May;76(5):1090-1099. doi: 10.1016/j.jhep.2021.12.038. Epub 2022 Jan 20. PMID 35066090
- [Derived] Simbrunner B, Semmler G, Stadlmann A, Scheiner B, Schwabl P, Paternostro R, Bucsics T, Bauer D, Eigenbauer E, Pinter M, Stattermayer AF, Quehenberger P, Marculescu R, Trauner M, Mandorfer M, Reiberger T. Vitamin A levels reflect disease severity and portal hypertension in patients with cirrhosis. Hepatol Int. 2020 Dec;14(6):1093-1103. doi: 10.1007/s12072-020-10112-3. Epub 2020 Dec 8. PMID 33289910
- [Derived] Costa D, Simbrunner B, Jachs M, Hartl L, Bauer D, Paternostro R, Schwabl P, Scheiner B, Stattermayer AF, Pinter M, Trauner M, Mandorfer M, Reiberger T. Systemic inflammation increases across distinct stages of advanced chronic liver disease and correlates with decompensation and mortality. J Hepatol. 2021 Apr;74(4):819-828. doi: 10.1016/j.jhep.2020.10.004. Epub 2020 Oct 16. PMID 33075344
- [Derived] Raeven P, Baron-Stefaniak J, Simbrunner B, Stadlmann A, Schwabl P, Scheiner B, Schaden E, Eigenbauer E, Quehenberger P, Mandorfer M, Baron DM, Reiberger T. Thromboelastometry in patients with advanced chronic liver disease stratified by severity of portal hypertension. Hepatol Int. 2020 Dec;14(6):1083-1092. doi: 10.1007/s12072-020-10093-3. Epub 2020 Sep 30. PMID 33000389
- [Derived] Simbrunner B, Marculescu R, Scheiner B, Schwabl P, Bucsics T, Stadlmann A, Bauer DJM, Paternostro R, Eigenbauer E, Pinter M, Stattermayer AF, Trauner M, Mandorfer M, Reiberger T. Non-invasive detection of portal hypertension by enhanced liver fibrosis score in patients with different aetiologies of advanced chronic liver disease. Liver Int. 2020 Jul;40(7):1713-1724. doi: 10.1111/liv.14498. Epub 2020 May 18. PMID 32358998